CLINICAL TRIAL: NCT06367218
Title: Opioid-Free Combined Anesthesia Under Spontaneous Breathing for Video-Assisted Thoracoscopic Surgery of Pulmonary Nodules: A Multicenter, Open-Label, Randomized Controlled, 2x2 Factorial Design Clinical Study
Brief Title: Opioid-Free Combined Anesthesia With Spontaneous Breathing for VATS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Hui Xu, professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S036
Record Dates: First submitted 2024-04-07; First posted 2024-04-16 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Video-assisted Thoracoscopic Lung Surgery；Anesthesia
MeSH Terms: interventions — Laryngeal Masks; Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- OSB (Experimental): Anesthesia was induced by intravenous injection of Sufentanil 0.1 µg/kg and propofol 2 mg /kg. The patient was placed with a laryngeal mask airway, connected to an anesthetic ventilator with spontaneous breathing mode. Anesthesia was maintained with propofol (5 mg/kg/h) and remifentanil (0.01 µg/kg/min) first, and then adjusted according to the depth of anesthesia.
  Paravertebral nerve blocks were performed at T4 and T6 levels with ropivacaine (0.5%, 10 ml) under ultrasound guidance. A mixture of 5 ml of 2% lidocaine and 5 ml of 0.5% ropivacaine was sprayed on the surface of the visceral pleura after thoracic cavity opening. The vagal and phrenic nerve trunks were blocked with 2 ml of the mixture.
  Interventions: Drug: opioid based strategy; Procedure: Laryngeal mask airway; Preserved spontaneous breathing
- KSB (Experimental): Anesthesia was induced by intravenous injection of Sufentanil 0.1 µg/kg and propofol 2 mg /kg. The patient was placed with a laryngeal mask airway, connected to an anesthetic ventilator with spontaneous breathing mode. Anesthesia was maintained with propofol (5 mg/kg/h) and remifentanil (0.01 µg/kg/min) first, and then adjusted according to the depth of anesthesia.
  Paravertebral nerve blocks were performed at T4 and T6 levels with ropivacaine (0.5%, 10 ml) under ultrasound guidance. A mixture of 5 ml of 2% lidocaine and 5 ml of 0.5% ropivacaine was sprayed on the surface of the visceral pleura after thoracic cavity opening. The vagal and phrenic nerve trunks were blocked with 2 ml of the mixture.
  Interventions: Drug: opioid-free strategy; Procedure: Laryngeal mask airway; Preserved spontaneous breathing
- OMV (Experimental): Anesthesia was induced by intravenous sufentanil injection of 0.5 μg/kg. Propofol 2 mg/kg and rocuronium 0.9 mg/kg were subsequently administered intravenously. After rocuronium took effect, double-lumen bronchial tube intubation was performed under the guidance of video laryngoscope, and fixed after the bronchoscopic examination, anesthesia ventilator was connected for mechanical ventilation, tidal volume was 6 mL/kg (ideal body weight), respiratory rate was 12-16 times /min, and end-expiratory partial pressure of carbon dioxide was maintained at 35-45 mmHg. Intraoperative anesthesia was maintained with initial intravenous pump of propofol (5 mg/kg/h) and remifentanil (0.1 μg/kg/min) first , and then adjusted according to the depth of anesthesia.
  Paravertebral nerve blocks were performed at T4 and T6 levels with ropivacaine (0.5%, 10 ml) under ultrasound guidance.
  Interventions: Drug: opioid based strategy; Procedure: Double lumen tracheal tube; Mechanical ventilation
- KMV (Experimental): Anesthesia was induced by intravenous injection of esketamine 0.5 mg/kg. Propofol 2 mg/kg and rocuronium 0.9 mg/kg were subsequently administered intravenously. After rocuronium took effect, double-chamber tracheal tube intubation was performed under the guidance of video laryngoscope, and fixed after the bronchoscopic examination, anesthesia ventilator was connected for mechanical ventilation, tidal volume was 6 mL/kg (ideal body weight), respiratory rate was 12-16 times /min, and end-expiratory partial pressure of carbon dioxide was maintained at 35-45 mmHg. Intraoperative anesthesia was maintained with the initial intravenous pump of propofol (5 mg/kg/h) and esketamine (0.5 mg/kg/h) first , and then adjusted according to the depth of anesthesia. Paravertebral nerve blocks were performed at T4 and T6 levels with ropivacaine (0.5%, 10 ml) under ultrasound guidance.
  Interventions: Drug: opioid-free strategy; Procedure: Double lumen tracheal tube; Mechanical ventilation

INTERVENTIONS:
Drug: opioid based strategy — Induction and maintenance of anesthesia with opioids
  Arms: OMV; OSB
Drug: opioid-free strategy — Esketamine was used for induction and maintenance of anesthesia
  Arms: KMV; KSB
Procedure: Laryngeal mask airway; Preserved spontaneous breathing — The patient used a laryngeal mask to maintain spontaneous breathing
  Arms: KSB; OSB
Procedure: Double lumen tracheal tube; Mechanical ventilation — The patient was mechanically ventilated using a double-lumen tracheal catheter
  Arms: KMV; OMV

SUMMARY:
Non-tracheal intubated combined anesthesia with preserved spontaneous breathing significantly enhances the quality and speed of recovery post-VATS for patients undergoing lung nodule surgery. The "opioid-sparing strategy," which substitutes ketamine for opioids during surgery, not only provides effective analgesia but also protects perioperative lung function and reasonably prevents the occurrence of opioid-related adverse reactions; it also reduces medical costs and shortens the average hospital stay. However, the degree of benefit to patients lacks high-level clinical evidence. This study aims to comprehensively assess the effect of opioid-free combined anesthesia with preserved spontaneous breathing for VATS lung nodule surgery on postoperative rapid recovery from multiple aspects including postoperative lung function and pulmonary complications, pain, gastrointestinal function, nausea/vomiting, cognitive function, and depression/anxiety, intending to expand the dataset and application prospects in this field, and increase feasibility experience.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized controlled, open-label, 2x2 factorial design trial involving two types of interventions: ventilation methods (2 levels: preserved spontaneous breathing, mechanical ventilation) and combined anesthesia methods (2 levels: opioid-free combined anesthesia, opioid-based combined anesthesia). To evaluate the clinical efficacy and safety of these two types of interventions, four parallel groups of patients undergoing video-assisted thoracoscopic surgery for pulmonary nodules under different anesthesia strategies were established: preserved spontaneous breathing and opioid-based combined anesthesia (OSB group), preserved spontaneous breathing and opioid-free combined anesthesia (KSB group), double-lumen endotracheal tube mechanical ventilation and opioid-based combined anesthesia (OMV group), and double-lumen endotracheal tube mechanical ventilation and opioid-free combined anesthesia (KMV group). This study will be conducted in the thoracic surgical centers of six hospitals in China, carried out by experienced senior anesthetists and thoracic surgeons. Patients undergoing anesthesia in this study will experience three observation phases. Phase 1 (perioperative phase, day 0 to day 2): Observing the lung function status and the occurrence of adverse events under different anesthesia plans during the perioperative period; Phase 2 (postoperative hospital stay, day 3 to day 7): Observing the lung function status and the occurrence of adverse events under different anesthesia plans during the hospital stay; Phase 3 (short-term follow-up, day 8 to day 30): Observing the lung function status and the occurrence of adverse events under different anesthesia plans during the short-term follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. ASA grades 1-2
2. Age > 18 years and < 70 years
3. Male or female patients
4. VATS pulmonary nodule operation is planned under general anesthesia
5. Voluntarily participate in the study and sign the informed consent

Exclusion Criteria:

1. Subject's operation is aborted
2. Serious adverse events, complications or special physiological changes during the perioperative period should not be continued
3. Expansion of surgical scope: resection of complex lung segment or complex lung lobectomy, thoracoscopic assisted small-incision surgery with enlarged incision, requiring pulmonary blood Tracheoplasty or bronchoplasty, partial pericardiectomy or conversion to thoracotomy
4. Those who need a second operation within a month
5. The patient or his/her guardian requests to withdraw on his/her own
6. Reasons why other researchers think the study needs to be discontinued

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Lung function 30 days after surgery | 30 days after surgery
  FEV1(% pred) at 30 days after thoracoscopic pulmonary nodule surgery.

SECONDARY OUTCOMES:
Intraoperative respiratory parameters | At the beginning of the operation, 30 minutes after the operation began, 1 hour, 2 hours, at the end of the operation
  Airway peak pressure
Intraoperative respiratory parameters | At the beginning of the operation, 30 minutes after the operation began, 1 hour, 2 hours, at the end of the operation
  oxygenation index (OI=PaO2/FiO2)
Intraoperative respiratory parameters | At the beginning of the operation, 30 minutes after the operation began, 1 hour, 2 hours, at the end of the operation
  alveolar arterial oxygen partial pressure difference (P(A-a)DO2)
Intraoperative respiratory parameters | At the beginning of the operation, 30 minutes after the operation began, 1 hour, 2 hours, at the end of the operation
  respiratory index (RI=P(A-a)DO2 /PaO2)
Intraoperative respiratory parameters | At the beginning of the operation, 30 minutes after the operation began, 1 hour, 2 hours, at the end of the operation
  dynamic lung compliance
Perioperative stage indicators | At the end of the operation
  Blood loss, intraoperative transfusion
Perioperative stage indicators | At the end of the operation
  operation time, anesthesia time, recovery time
Postoperative pain | Six hours, 24 hours, 48 hours after surgery
  Postoperative pain (numerical rating scale (NRS))
Postoperative Lung function | 1, 3, 5 days after surgery
  FVC, FEV1, FEV1 (% pred)
Postoperative Lung function | 1, 3, 5 days after surgery
  Copd Patient Self-Assessment Test (CAT)，Scores range from 0 to 40, with ≥10 indicating the need for medical intervention.
Postoperative pulmonary complications | 1, 3, 5 days after surgery
  european perioperative clinical outcome (EPCO)
Postoperative gastrointestinal function | Six hours, 24 hours, 48 hours after surgery
  Intake, Feeling nauseated, Emesis, Exam, and Duration of symptoms scoring system, I-FEED，0 ~ 2 points, normal; 3 ~ 5 scores, postoperative gastrointestinal functional intolerance; ≥6 points, POGD.
Postoperative depression/anxiety | Before surgery, 2 days after surgery
  (hospital anxiety and depression scale, HADS) scale score，Anxiety and depression were divided into two subscales: 0-7 was negative; 8-10 is mild; 11-14 divided into moderate; 15 to 21 is classified as severe
Postoperative cognitive function | Before surgery, 1 day after surgery, 3 days after surgery
  (mini-mental state examination, MMSE) scale score，The maximum score is 30 points. The classification of dementia is related to the level of education, so if the elderly are illiterate and less than 17 points, primary school and less than 20 points, secondary school and above less than 24 points, then dementia.
Time of first exercise after surgery | From the end of surgery，Until the first time of off-bed activity
  objective parameters included stable vital signs, no obvious bleeding tendency, NRS score less than 5 points
The 6-minute walking experiment | 30 days after surgery.
  Measure the distance covered by an individual walking for 6 minutes at the highest speed
Length of stay | From date of surgery Until the date of discharge or death
  The number of days spent in the hospital from the end of surgery until discharge or death
Quality of life measurement | the date of discharge，and Thirty days after surgery
  Use a WHOQOL-BREF scale rating to evaluate quality of life
Intraoperative circulation parameters | At the beginning of the operation, 30 minutes after the operation began, 1 hour, 2 hours, at the end of the operation
  Blood pressure
Intraoperative circulation parameters | At the beginning of the operation, 30 minutes after the operation began, 1 hour, 2 hours, at the end of the operation
  heart rate
Intraoperative circulation parameters | At the beginning of the operation, 30 minutes after the operation began, 1 hour, 2 hours, at the end of the operation
  pulse oxygen saturation
Intraoperative circulation parameters | At the beginning of the operation, 30 minutes after the operation began, 1 hour, 2 hours, at the end of the operation
  anesthesia depth index
Intraoperative circulation parameters | At the beginning of the operation, 30 minutes after the operation began, 1 hour, 2 hours, at the end of the operation
  body temperature
Intraoperative circulation parameters | At the beginning of the operation, 30 minutes after the operation began, 1 hour, 2 hours, at the end of the operation
  urine volume

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No